CLINICAL TRIAL: NCT03945240
Title: Evaluating Different Low-level Laser Therapies to Treat Neck Pain in Air Force Pilots and Flight Crew
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find qualified subjects and lack of funding
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20190105H
Record Dates: First submitted 2019-05-01; First posted 2019-05-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Pinnacle, lower dosimetry parameters) (Experimental): Utilize the Pinnacle Series Laser by Aspen Laser Systems to apply LLLT
  Interventions: Procedure: Group 1 -- using Pinnacle Series Laser Device
- Group 2 (Pinnacle, higher dosimetry parameters) (Experimental): Utilize the Pinnacle Series Laser by Aspen Laser Systems to apply LLLT
  Interventions: Procedure: Group 2 -- using Pinnacle Series Laser Device
- Group 3 (Phoenix) (Experimental): Utilizing the Phoenix Thera-Lase by Phoenix Thera-Lase Systems, we will apply LLT.
  Interventions: Procedure: Group 3 -- using Phoenix Thera-Lase Device

INTERVENTIONS:
Procedure: Group 1 -- using Pinnacle Series Laser Device — Utilizing the Pinnacle Series Laser by Aspen Laser Systems, investigators will apply 635-780nm, 10 mW cw, ~ 5-105 J/cm2 at the following time and mW intervals. The beam will be applied at 12 application patterns equidistant and parallel to each other. Each application point will be treated for the timeframes referenced below:
  * Subgroup 1: 10 minutes at 5 mW
  * Subgroup 2: 10 minutes at 15 mW
  * Subgroup 3: 10 minutes at 32 mW
  * Subgroup 4: 15 minutes at 5 mW
  * Subgroup 5: 15 minutes at 15 mW
  * Subgroup 6: 15 minutes at 32 mW
  Arms: Group 1 (Pinnacle, lower dosimetry parameters)
Procedure: Group 2 -- using Pinnacle Series Laser Device — Utilizing the Pinnacle Series Laser by Aspen Laser Systems, we will apply 830nm, 30- 50mW cw, ~ 1-20 J/cm2 at the following time and mW intervals. The beam will be applied at 12 application patterns equidistant and parallel to each other. Each application point will be treated for the timeframes referenced below:
  * Subgroup 1: 10 minutes at 5 mW
  * Subgroup 2: 10 minutes at 15 mW
  * Subgroup 3: 10 minutes at 32 mW
  * Subgroup 4: 15 minutes at 5 mW
  * Subgroup 5: 15 minutes at 15 mW
  * Subgroup 6: 15 minutes at 32 mW
  Arms: Group 2 (Pinnacle, higher dosimetry parameters)
Procedure: Group 3 -- using Phoenix Thera-Lase Device — Utilizing the Phoenix Thera-Lase by Phoenix Thera-Lase Systems, we will apply 904nm, 40mW (pulsed) @10000Hz, ~ 4-18 J/cm2 at the following time and mW intervals. The beam will be applied at 12 application patterns equidistant and parallel to each other. Each application point will be treated for the timeframes referenced below:
  * Subgroup 1: 10 minutes at 5 mW
  * Subgroup 2: 10 minutes at 15 mW
  * Subgroup 3: 10 minutes at 32 mW
  * Subgroup 4: 15 minutes at 5 mW
  * Subgroup 5: 15 minutes at 15 mW
  * Subgroup 6: 15 minutes at 32 mW
  Arms: Group 3 (Phoenix)

SUMMARY:
Determine the most effective and efficient treatment protocols for treating neck pain with LLLT.

DETAILED DESCRIPTION:
The purpose of this study is to identify what are the most effective low level laser therapy (LLLT) dosimetry parameters when treating pilots and navigators complaining of flight related neck pain.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty US Air Force pilots or onboard navigators, aged 18- 62 years of age
* maintain operational flight status at enrollment or within the last 6 months
* History of neck pain for a period of more than two months
* Score on the Neck Disability Index ranging from 15-24
* No physiotherapy or local injection in 3 months before starting the study

Exclusion Criteria:

* pregnant
* major surgery or trauma in the previous 3 months
* unstable cervical spine
* cervical radiculopathy
* rheumatoid arthritis
* open wound over neck
* pace-maker or defibrillator implantation
* overt neuropathic pain or radiation pain
* inability to express pain or quality of life.
* history of neurological disorders
* medical diagnosis of fibromyalgia; systemic disease

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Number of grounding days from flying due to neck pain -- Interval Variable | Record during screening visit
  Number of grounding days from flying due to neck pain -- Interval Variable
Change in Neck Disability Index (NDI) | visit 0 (screening visit), visit 1 (day 1), visit 10 (day 10)
  The NDI assessing functional capacity, has 10 parts, which evaluate pain intensity, personal care, lifting objects, reading, headache, concentration, work, driving, sleeping, and recreation. NDI scores, ranging from 0-50, may be doubled and also expressed as a percentage of function on a scale of 0-100%; thereby allowing the measure to be treated as an interval variable. It has also been categorized into 5 ordinal measurements, which are shown below with corresponding score and percentage measurements:
  * NDI Score 0-4 (0-8%) is total capacity (no disability)
  * NDI Score 5-14 (10-28%) is mild incapacity (mild disability)
  * NDI Score 15-24 (30-48%) is mild incapacity (moderate disability)
  * NDI Score 25-34 (50-64%) is serious capacity (severe disability)
  * NDI Score 35-50 (70-100%) is severe incapacity (complete disability)
Change in Defense and Veterans Pain Rating Scale (DVPRS) | visit 0 (screening visit), visit 1 (day 1), visit 10 (day 10)
  The Defense and Veterans Pain Rating Scale is an assessment tool that utilizes a numerical rating scale, enhanced by functional word descriptors, color coding, and graphical facial expressions to evaluate a patient's self-reported pain levels.
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.

SECONDARY OUTCOMES:
Change in Interleukin 2 Receptor (CD25) Soluble Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 2 Receptor (CD25) Soluble
  Standard curve range: 4.25-17400 pg/mL
Change in Interleukin 12 biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 12
  Standard curve range: 1.56-6400 pg/mL
Change in Interleukin 4 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 4
  Standard curve range: 9.35-38300 pg/mL
Change in Interleukin 5 biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 5
  Standard curve range: 6.52-26700 pg/mL
Change in Interleukin 10 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 10
  Standard curve range: 2.49-10200 pg/mL
Change in Interleukin 13 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 13
  Standard curve range: 3.27-13400 pg/mL
Change in Interleukin 1 beta Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 1 beta
  Standard curve range: 2.39-9800 pg/mL
Change in Interleukin 6 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 6
  Standard curve range: 6.74-27600 pg/mL
Change in Interleukin 8 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 8
  Standard curve range: 2.38-9750 pg/mL
Change in Tumor Necrosis Factor - alpha Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Tumor Necrosis Factor - alpha
  Standard curve range: 6.42-26300 pg/mL
Change in Interleukin 2 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 2
  Standard curve range: 4.25-17400 pg/mL
Change in Interleukin 17 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  Interleukin 17
  Standard curve range: 2.22-9100 pg/mL
Change in cyclooxygenase (COX-2 Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  cyclooxygenase (COX-2)
  Standard curve range: 7.5 U/ml - 60 U/ml
Change in cortisol Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  cortisol
  * Standard curve range: cortisol will be compared to normal reference range for the time the blood is drawn, which is noted on lab report
  * 8AM sample using the new assays is 10 to 50 picograms per milliliter (pg/ml); levels are usually less than 20 pg/ml at 4 PM and less than 5-10 pg/ml at midnight.
Change in substance P Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  substance P
  Standard curve range: N/A, values from day 0 time will be compared with day 10 values
Change in C-reactive protein Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  C-reactive protein
  Standard curve range: 3 mg/L-10 mg/L
Change in alpha-1 antitrypsin Biomarker Levels | day 0 (pre-treatment), day 10 (post-treatment)
  Phlebotomists will draw 750 uL into 3 separate cryovials on two separate occasions.
  alpha-1 antitrypsin
  Standard curve range: 100-300 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Principal Investigator — US Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Hamalainen O, Heinijoki H, Vanharanta H. Neck training and +Gz-related neck pain: a preliminary study. Mil Med. 1998 Oct;163(10):707-8. PMID 9795549
- [Background] Harrison MF, Neary JP, Albert WJ, Kuruganti U, Croll JC, Chancey VC, Bumgardner BA. Measuring neuromuscular fatigue in cervical spinal musculature of military helicopter aircrew. Mil Med. 2009 Nov;174(11):1183-9. doi: 10.7205/milmed-d-00-7409. PMID 19960827
- [Background] Salmon DM, Harrison MF, Neary JP. Neck pain in military helicopter aircrew and the role of exercise therapy. Aviat Space Environ Med. 2011 Oct;82(10):978-87. doi: 10.3357/asem.2841.2011. PMID 21961403
- [Background] (2018) International Association for the Study of Pain : Neck pain.
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Attal N, Lanteri-Minet M, Laurent B, Fermanian J, Bouhassira D. The specific disease burden of neuropathic pain: results of a French nationwide survey. Pain. 2011 Dec;152(12):2836-2843. doi: 10.1016/j.pain.2011.09.014. Epub 2011 Oct 20. PMID 22019149
- [Background] Torrance N, Ferguson JA, Afolabi E, Bennett MI, Serpell MG, Dunn KM, Smith BH. Neuropathic pain in the community: more under-treated than refractory? Pain. 2013 May;154(5):690-699. doi: 10.1016/j.pain.2012.12.022. Epub 2013 Jan 23. PMID 23485369
- [Background] Mester E, Ludany G, Sellyei M, Szende B, Gyenes G, Tota GJ. [Studies on the inhibiting and activating effects of laser beams]. Langenbecks Arch Chir. 1968;322:1022-7. doi: 10.1007/BF02453990. No abstract available. German. PMID 5758676
- [Background] Avci P, Gupta A, Sadasivam M, Vecchio D, Pam Z, Pam N, Hamblin MR. Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg. 2013 Mar;32(1):41-52. PMID 24049929
- [Background] (2018) North American Association for Photobiomodulation Therapy.
- [Background] Guarini D, Gracia B, Ramirez-Lobos V, Noguera-Pantoja A, Sole-Ventura P. Laser Biophotomodulation in Patients with Neurosensory Disturbance of the Inferior Alveolar Nerve After Sagittal Split Ramus Osteotomy: A 2-Year Follow-Up Study. Photomed Laser Surg. 2018 Jan;36(1):3-9. doi: 10.1089/pho.2017.4312. Epub 2017 Oct 12. PMID 29022844
- [Background] Chow RT, Heller GZ, Barnsley L. The effect of 300 mW, 830 nm laser on chronic neck pain: a double-blind, randomized, placebo-controlled study. Pain. 2006 Sep;124(1-2):201-10. doi: 10.1016/j.pain.2006.05.018. Epub 2006 Jun 27. PMID 16806710
- [Background] Enwemeka CS, Parker JC, Dowdy DS, Harkness EE, Sanford LE, Woodruff LD. The efficacy of low-power lasers in tissue repair and pain control: a meta-analysis study. Photomed Laser Surg. 2004 Aug;22(4):323-9. doi: 10.1089/pho.2004.22.323. PMID 15345176
- [Background] Carrasco TG, Guerisoli LD, Guerisoli DM, Mazzetto MO. Evaluation of low intensity laser therapy in myofascial pain syndrome. Cranio. 2009 Oct;27(4):243-7. doi: 10.1179/crn.2009.035. PMID 19891258
- [Background] Olavi A, Pekka R, Pertti K, Pekka P. Effects of the infrared laser therapy at treated and non-treated trigger points. Acupunct Electrother Res. 1989;14(1):9-14. doi: 10.3727/036012989816358560. PMID 2568075
- [Background] Graham N, Gross AR, Carlesso LC, Santaguida PL, Macdermid JC, Walton D, Ho E; ICON. An ICON Overview on Physical Modalities for Neck Pain and Associated Disorders. Open Orthop J. 2013 Sep 20;7:440-60. doi: 10.2174/1874325001307010440. eCollection 2013. PMID 24155804
- [Background] Ceccherelli F, Altafini L, Lo Castro G, Avila A, Ambrosio F, Giron GP. Diode laser in cervical myofascial pain: a double-blind study versus placebo. Clin J Pain. 1989 Dec;5(4):301-4. doi: 10.1097/00002508-198912000-00005. PMID 2520419
- [Background] Ozdemir F, Birtane M, Kokino S. The clinical efficacy of low-power laser therapy on pain and function in cervical osteoarthritis. Clin Rheumatol. 2001;20(3):181-4. doi: 10.1007/s100670170061. PMID 11434469
- [Background] Konstantinovic LM, Cutovic MR, Milovanovic AN, Jovic SJ, Dragin AS, Letic MDj, Miler VM. Low-level laser therapy for acute neck pain with radiculopathy: a double-blind placebo-controlled randomized study. Pain Med. 2010 Aug;11(8):1169-78. doi: 10.1111/j.1526-4637.2010.00907.x. PMID 20704667
- [Background] Gur A, Sarac AJ, Cevik R, Altindag O, Sarac S. Efficacy of 904 nm gallium arsenide low level laser therapy in the management of chronic myofascial pain in the neck: a double-blind and randomize-controlled trial. Lasers Surg Med. 2004;35(3):229-35. doi: 10.1002/lsm.20082. PMID 15389743
- [Background] Ilbuldu E, Cakmak A, Disci R, Aydin R. Comparison of laser, dry needling, and placebo laser treatments in myofascial pain syndrome. Photomed Laser Surg. 2004 Aug;22(4):306-11. doi: 10.1089/pho.2004.22.306. PMID 15345173
- [Background] Hakguder A, Birtane M, Gurcan S, Kokino S, Turan FN. Efficacy of low level laser therapy in myofascial pain syndrome: an algometric and thermographic evaluation. Lasers Surg Med. 2003;33(5):339-43. doi: 10.1002/lsm.10241. PMID 14677161
- [Background] Woodruff LD, Bounkeo JM, Brannon WM, Dawes KS, Barham CD, Waddell DL, Enwemeka CS. The efficacy of laser therapy in wound repair: a meta-analysis of the literature. Photomed Laser Surg. 2004 Jun;22(3):241-7. doi: 10.1089/1549541041438623. PMID 15315732
- [Background] Huang YY, Chen AC, Carroll JD, Hamblin MR. Biphasic dose response in low level light therapy. Dose Response. 2009 Sep 1;7(4):358-83. doi: 10.2203/dose-response.09-027.Hamblin. PMID 20011653
- [Background] Huang YY, Sharma SK, Carroll J, Hamblin MR. Biphasic dose response in low level light therapy - an update. Dose Response. 2011;9(4):602-18. doi: 10.2203/dose-response.11-009.Hamblin. Epub 2011 Sep 2. PMID 22461763
- [Background] Huang YY, Nagata K, Tedford CE, McCarthy T, Hamblin MR. Low-level laser therapy (LLLT) reduces oxidative stress in primary cortical neurons in vitro. J Biophotonics. 2013 Oct;6(10):829-38. doi: 10.1002/jbio.201200157. Epub 2012 Dec 27. PMID 23281261
- [Background] Huang YY, Nagata K, Tedford CE, Hamblin MR. Low-level laser therapy (810 nm) protects primary cortical neurons against excitotoxicity in vitro. J Biophotonics. 2014 Aug;7(8):656-64. doi: 10.1002/jbio.201300125. Epub 2013 Oct 15. PMID 24127337